CLINICAL TRIAL: NCT02502396
Title: Retrospective Study: Rivaroxaban Utilization for Treatment and Prevention of Thromboembolism in Cancer Patients: Experience at a Comprehensive Cancer Center
Brief Title: Rivaroxaban Utilization for Treatment and Prevention of Thromboembolism in Cancer Patients: Experience at a Comprehensive Cancer Center
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: PA14-1027
Record Dates: First submitted 2015-07-14; First posted 2015-07-20 (Estimated); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Cancer; Deep-vein Thrombosis of the Lower and Upper Extremities; Pulmonary Embolism; Non-valvular Atrial Fibrillation
Keywords: Cancer; Deep-vein thrombosis of the lower and upper extremities; Pulmonary embolism; Non-valvular atrial fibrillation; Chart review; VTE; NVAF; Rivaroxaban
MeSH Terms: conditions — Neoplasms; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chart Review - Patterns of Rivaroxaban Usage: Retrospective chart review study to evaluate Rivaroxaban's utilization in cancer patients for venous-thromboembolism (VTE) or non-valvular atrial fibrillation (NVAF).
  Interventions: Other: Retrospective Chart Review

INTERVENTIONS:
Other: Retrospective Chart Review — Retrospective chart review study to evaluate Rivaroxaban's utilization in cancer patients for venous-thromboembolism (VTE) or non-valvular atrial fibrillation (NVAF). Study conducted from from January 1, 2012 to November 7, 2016 at MD Anderson Cancer Center in Houston, Texas.

SUMMARY:
The primary objective of this study is to evaluate the practice patterns of rivaroxaban usage invenous-thromboembolism (VTE) and non-valvular atrial fibrillation (NVAF) in cancer patients.

The secondary objectives are to evaluate outcomes such as recurrent VTE, stroke and bleeding for cancer patients on rivaroxaban.

DETAILED DESCRIPTION:
This retrospective descriptive study will review charts of approximately 375 cancer patients prescribed rivaroxaban from January 1, 2012 to November 7, 2016 at UT MDACC for NVAF or patients that had prior VTE and diagnosis of cancer. The list of patients prescribed rivaroxaban during the study period will be obtained from Pharmacy Informatics. We will review the eligibility of all patients on the pharmacy list who were prescribed rivaroxaban during the study time-frame. The eligible patients who meet inclusion/exclusion criteria will be identified. All available data concerning demographic, clinical parameters and rivaroxaban usage will be collected for eligible patients from Pharmacy Informatics, CS, Laboratory Informatics, and Clinical Informatics Databases.

The variables of interest include demographic information, clinical parameters (tumor type, extent of disease, clinical exam findings, and presence of comorbidities, diagnostic assessments, and treatment interventions), reason for rivaroxaban discontinuation and outcomes. The confidentiality of all patient-specific data will be maintained. By using Pharmacy Informatics and CS, we can capture most of patients prescribed rivaroxaban at the UT MDACC.This is a descriptive study and the final sample size will depend on available records for chart review from 01/01/2012 to 11/07/2016.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: patient must be ≥ 18 years.
2. Male and female patients will be eligible for enrollment.
3. Patients diagnosed with deep-vein thrombosis of the lower and upper extremities, pulmonary embolism or both or with non-valvular atrial fibrillation.
4. Patients must have active malignancy defined as a diagnosis of cancer (excluding basal cell squamous cell carcinoma of the skin) within six months before enrollment, have received any treatment for cancer within the previous six months or have documented recurrent or metastatic cancer .

Exclusion Criteria:

1. Patients who are on hemodialysis
2. Patients with valvular heart disease (using a coexisting prosthetic heart valve or have a hemodynamically significant valve disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients with venous-thromboembolism (VTE) or non-valvular atrial fibrillation (NVAF) The University of Texas MD Anderson Cancer Center in Houston, Texas
Sampling Method: Probability Sample
Enrollment: 265 (Actual)
Dates: Start 2015-09-28 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Chart Review of Usage Pattern of Rivaroxaban in Participants with Cancer and Invenous-Thromboembolism (VTE) at MD Anderson Cancer Center | 1 year
  Proportion (95% confidence interval (CI)) of cancer patients who were on rivaroxaban with indication of VTE obtained among cancer patients who were on rivaroxaban.
  Analyses made among patients with VTE summarizing practice patterns of rivaroxaban by means, SDs, and ranges for continuous variables (e.g. platelet counts before a procedure) and the counts and percentages for categorical variables (e.g. stopping rivaroxaban before a procedure, stopping rivaroxaban when the platelets dropped < 50K, adjusting rivaroxaban dose when the platelets dropped < 50K, restarting rivaroxaban after it stopped).
Chart Review of Usage Pattern of Rivaroxaban in Participants with Cancer and Non-Valvular Atrial Fibrillation (NVAF) at MD Anderson Cancer Center | 1 year
  Proportion (95% confidence interval (CI)) of cancer patients who were on rivaroxaban with indication of NVAF obtained among cancer patients who were on rivaroxaban.
  Analyses made among patients with NVAF summarizing practice patterns of rivaroxaban by means, SDs, and ranges for continuous variables (e.g. platelet counts before a procedure) and the counts and percentages for categorical variables (e.g. stopping rivaroxaban before a procedure, stopping rivaroxaban when the platelets dropped < 50K, adjusting rivaroxaban dose when the platelets dropped < 50K, restarting rivaroxaban after it stopped).

SECONDARY OUTCOMES:
Chart Review of Stroke Outcome Evaluation of Rivaroxaban in Cancer Participants with Invenous-Thromboembolism (VTE) at MD Anderson Cancer Center | 1 year
  Proportions of patients with recurrent stroke along with 95% CIs, estimated among patients with VTE . SAS 9.4 (SAS Institute INC, Cary, NC) used for data analysis.
Chart Review of Bleeding Outcome Evaluation of Rivaroxaban in Cancer Participants with Invenous-Thromboembolism (VTE) at MD Anderson Cancer Center | 1 year
  Proportions of patients with recurrent bleeding, along with 95% CIs, estimated among patients with VTE. SAS 9.4 (SAS Institute INC, Cary, NC) used for data analysis.
Chart Review of Stroke Outcome Evaluation of Rivaroxaban in Cancer Participants with Non-Valvular Atrial Fibrillation (NVAF) at MD Anderson Cancer Center | 1 year
  Proportions of patients with recurrent NVAF along with 95% CIs, estimated among patients with NVAF. SAS 9.4 (SAS Institute INC, Cary, NC) used for data analysis.
Chart Review of Bleeding Outcome Evaluation of Rivaroxaban in Cancer Participants with Non-Valvular Atrial Fibrillation (NVAF) at MD Anderson Cancer Center | 1 year
  Proportions of patients with recurrent bleeding, along with 95% CIs, estimated among patients with NVAF. SAS 9.4 (SAS Institute INC, Cary, NC) used for data analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Escalante, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org